CLINICAL TRIAL: NCT05303168
Title: Prevalence and Impact of SARS-CoV-2 Infection on Maternal and Infant Health in African Populations (MA-CoV)
Brief Title: Prevalence and Impact of COVID-19 on Maternal and Infant Health in African Populations
Acronym: MA-CoV
Status: Completed | Type: Observational
Sponsor: Barcelona Institute for Global Health (Other)
Collaborators: Centre de Recherche Médicale de Lambaréné (Other); Centro de Investigação em Saúde de Manhiça (Other); Universität Tübingen (Other); Bernhard Nocht Institute for Tropical Medicine (Other Government)
Responsible Party: Sponsor
Other Study IDs: RIA2020EF-2956
Record Dates: First submitted 2022-03-10; First posted 2022-03-31 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: SARS-CoV2 Infection; COVID-19
Keywords: SARS-CoV-2; COVID-19; Pregnancy; Perinatal; Sub-Saharan Africa
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is growing evidence that COVID-19 threatens maternal and perinatal health. Pregnant women are at higher risk of severe complications (severe pneumonia, hospitalizations, intensive care unit admission, invasive mechanical ventilation, extracorporeal membrane oxygenation) and death compared to age-matched non-pregnant women. On the other hand, the number of confirmed COVID-19 cases reported in sub-Saharan Africa (SSA) continues to increase, where the highest maternal mortality rates in the world are registered. The World Health Organization (WHO) estimates that this region alone accounted for roughly two-thirds (196 000) of all maternal deaths in 2017, which among other reasons is explained by the inequalities in access to quality antenatal care (ANC) services and the low numbers of skilled health workers in the region. The spread of SARS-CoV-2 in SSA is threatening the already fragile health services, affecting mainly the most vulnerable populations such as pregnant women.

This project aims to describe the burden and effects of SARS-CoV-2 infection during pregnancy in women living in malaria endemic areas and high prevalence of HIV infection. Pregnant women attending ANC clinics in selected sites from Libreville and Lambaréné (Gabon) and Manhiça (Mozambique) will be enrolled in a cohort study to determine the frequency of SARS-CoV-2 infection and COVID-19 during pregnancy and its effects on maternal and neonatal health. Participants will be tested for SARS-CoV-2 infection whenever reporting respiratory symptoms suggestive of COVID-19 during routine ANC follow-up and six weeks after the end of pregnancy. The presence of antibodies (IgG/IgM) against SARS CoV-2 in blood samples will be determined. The clinical presentation of COVID-19 in pregnancy will be also characterised, and the incidence of infection during pregnancy and the risk factors of maternal and neonatal morbidity and mortality associated with SARS-CoV-2 infection and the frequency of mother- to- child transmission of SARS-CoV-2 will be assessed.

The findings of this project will contribute to the understanding of the impact of SARS-CoV-2 and COVID-19 among pregnant women living in SSA countries where malaria and HIV infections are highly prevalent.

ELIGIBILITY:
Inclusion Criteria:

* Permanent resident in the study area
* Agreement to deliver in the study site's maternity(ies) wards

Exclusion Criteria:

* Planning to move out the study area in the following 7 months from enrolment

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be pregnant women of all gravidities attending the antenatal care (ANC) clinics of the study sites in Gabon and Mozambique.
  Inclusion of legal minors will follow local national guidelines from Gabon and Mozambique. If the woman is under the legal age of maturity, she will sign the assent form and a legal guardian of the woman will sign the informed consent form.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of antibodies (Ig G and/or Ig M positive) against SARS-CoV-2 among pregnant women at delivery | 7 months

SECONDARY OUTCOMES:
Incidence of SARS-CoV-2 infection during pregnancy | 7 months
Maternal and neonatal morbidity due to SARS-CoV-2 infection during pregnancy | 7 months
Maternal and neonatal mortality due to SARS-CoV-2 infection during pregnancy | 7 months
Prevalence of pregnancy and perinatal adverse outcomes | 7 months
Rate of vertical transmission of SARS-CoV-2 from infected mothers to their offspring, during the prenatal and perinatal period | 7 months
CD4 cell counts | 7 months
HIV viral load | 7 months
Frequency of malaria parasitaemia at delivery (from maternal sample collected at delivery) | 7 months

CONTACTS AND LOCATIONS:
Locations (2):
- Centre de Recherches Médicales de Lambaréné (CERMEL), Lambaréné, Gabon
- Centro de Investigação em Saúde de Manhiça (CISM), Manhiça, Mozambique

REFERENCES:
- [Background] Figueroa-Romero A, Mendes A, Mombo-Ngoma G, Mischlinger J, Esen M, Vogler M, Mazuze M, Mombo-Nzamba L, Mbadinga B, Sanz S, Ramharter M, Saute F, Nhampossa T, Menendez C, Gonzalez R. Prevalence and impact of SARS-CoV-2 infection on maternal and infant health in African populations: protocol of a multicentre prospective cohort study (MA-CoV project). BMJ Open. 2023 May 22;13(5):e067083. doi: 10.1136/bmjopen-2022-067083. PMID 37217271
- [Result] Gonzalez R, Nhampossa T, Figueroa-Romero A, Mendes A, Mazuze M, Garcia-Otero L, Sevene E, Piqueras M, Egri N, Bedini JL, Saute F, Menendez C. SARS-CoV-2 Seropositivity and HIV Viral Load Among Mozambican Pregnant Women. J Acquir Immune Defic Syndr. 2023 Feb 1;92(2):115-121. doi: 10.1097/QAI.0000000000003120. Epub 2022 Oct 26. PMID 36287578